CLINICAL TRIAL: NCT00983203
Title: Acute Comfort and Haze Profile of FID 114657
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: C-09-014
Record Dates: First submitted 2009-09-23; First posted 2009-09-24 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-01

CONDITIONS: Dry Eye
Keywords: Dry eye; artificial tears
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- FID 114657 (Experimental): FID 114657
  Interventions: Other: FID 114657 ORB Preserved Ocular Emulsion
- Soothe XP Lubricant Eye Drops (Active Comparator): Soothe XP Lubricant Eye Drops
  Interventions: Other: Soothe XP Lubricant Eye Drops

INTERVENTIONS:
Other: FID 114657 ORB Preserved Ocular Emulsion — 1 drop OU
  Arms: FID 114657
Other: Soothe XP Lubricant Eye Drops — 1 drop OU
  Arms: Soothe XP Lubricant Eye Drops

SUMMARY:
The purpose of this study is to describe the acute comfort and haze profile of FID 114657 in dry eye patients.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of dry eye

Exclusion Criteria:

* Must not have worn contact lenses for 1 week preceding enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-07; Primary Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Drop comfort upon instillation | Upon instillation